CLINICAL TRIAL: NCT05711641
Title: Action of Intra-auricular Topical Lidocaine on Tinnitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Ricardo Ferreira Bento, PhD, Professor of Otorhinolaringology Department of Faculdade de Medicina da Universidade de São Paulo, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 5562868
Record Dates: First submitted 2023-01-21; First posted 2023-02-03 (Actual); Results first posted 2024-08-30 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Tinnitus, Subjective
Keywords: tinnitus; lidocaine; tinnitus treatment; tinnitus diagnosis; tinnitus suppression
MeSH Terms: conditions — Tinnitus | interventions — Lidocaine; compact-colony-forming active substance

STUDY DESIGN:
Intervention Model Description: All patients will receive both lidocaine and placebo at an interval of 15 days and the order of application of the substances is randomized.
Who Masked: Participant, Investigator
Masking Description: This is a double blind study. The substances are produced by the same handling pharmacy and delivered in identical vials, only with the information: substance 1 and substance 2.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lidocaine 10% (Experimental): The patient is instructed to lie down in lateral decubitus, with the ear in study facing upwards and 10% lidocaine is applied to the external auditory canal, using an eyedropper, until its complete filling (approximate average of 2ml).
  Interventions: Drug: Lidocaine 10 MG/ML
- Placebo (Placebo Comparator): The patient is instructed to lie down in lateral decubitus, with the ear in study facing upwards and distilled water is applied to the external auditory canal, using an eyedropper, until its complete filling (approximate average of 2ml).
  Interventions: Drug: Distilled water

INTERVENTIONS:
Drug: Lidocaine 10 MG/ML — Application of 10% topical lidocaine in the external auditory canal of tinnitus patients.
  Other Names: Active substance
  Arms: Lidocaine 10%
Drug: Distilled water — Application of distilled water in the external auditory canal of tinnitus patients.
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The main objective of this clinical trial placebo controled is to evaluate the action of intraauricular topical lidocaine on tinnitus.

The question to be answered is whether lidocaine is superior to placebo (distilled water) in reducing tinnitus intensity when applied topically within the external auditory canal.

Tinnitus intensity will be measured using the visual analog scale and acuphenometry before and after lidocaine or placebo application.

DETAILED DESCRIPTION:
Adult patients who have had continuous, uni or bilateral tinnitus, for at least 6 months are being evaluated. Exclusion criteria are: otological infection, tympanic membrane perforation, anatomical alteration of the external ear, pulsatile tinnitus, objective tinnitus, known allergy to lidocaine or other topical anesthetic and pregnancy All patients receive both lidocaine and placebo at an interval of 15 days and the order of application of the substances is randomized. Only one ear receives the medications and side is defined by the higher intensity of tinnitus, or through draw in the case of symmetrical tinnitus.

The patient is instructed to lie in lateral decubitus, with the ear under study facing upwards and the substances are applied by filling the external auditory canal with lidocaine or distilled water for 5 min. Tinnitus intensity is measured (acuphenometry and VAS) before and after substance application and the variation is compared between lidocaine and placebo.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who have had continuous, uni or bilateral tinnitus, for at least 6 months

Exclusion Criteria:

* Otological infection
* Tympanic membrane perforation
* Anatomical alteration of the external ear
* Pulsatile tinnitus
* Objective tinnitus
* Known allergy to lidocaine or other topical anesthetic and pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-09-02 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo F Bento, Principal Investigator — University of Sao Paulo
Locations (1):
- Faculdade de Medicina da Universidade de São Paulo, São Paulo, Brazil

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The selected subjects were patients of an otolaryngology center who sought care for tinnitus complaints between April 7, 2021, to April 6, 2022. Of them, 113 patients met the inclusion criteria, and none of the exclusion criteria, and were invited to participate in the study through WhatsApp contact. Thirty-three patients responded and attended the initial appointment, one was excluded for having only pulsatile tinnitus on the day of the appointment. Thirty two were enrolled.
Pre-assignment Details: Thirty-three patients responded and attended the initial appointment, one was excluded for having only pulsatile tinnitus on the day of the appointment.
  Thirty-two patients started the study, being divided into study group (n=16) or placebo (n=16) through randomization. Each patient was their own control because this was a crossover study with an interval of 2 weeks between each evaluation.
Groups:
- Lidocaine 10%, Then Placebo: The patients underwent a single, topical intraauricular dose of lidocaine 10%. After a two-week washout, the same subjects underwent a single dose, topical intraauricular distilled water (placebo).
- Placebo, Then lidocaíne 10%: The patients underwent a single, topical intraauricular dose of distilled water (placebo). After a two-week washout, the same subjects underwent a single dose, topical intra-auricular lidocaine 10%.
Period: First Intervention (Single Dose)
Arm/Group | Lidocaine 10%, Then Placebo | Placebo, Then lidocaíne 10%
Started | 16 (Sixteen patients (16) were randomly assigned to the lidocaine then placebo group. The patients received a single application of 10% lidocaine via intraauricular contact.) | 16 (Sixteen patients were randomly assigned to the placebo then lidocaine group. The patients received a single application of distilled water via intraauricular contact.)
Completed | 16 | 16
Not Completed | 0 | 0
Period: Washout (2 Weeks)
Arm/Group | Lidocaine 10%, Then Placebo | Placebo, Then lidocaíne 10%
Started | 16 | 16
Completed | 14 | 15
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 2 | 1
Period: Second Intervention (Single Dose)
Arm/Group | Lidocaine 10%, Then Placebo | Placebo, Then lidocaíne 10%
Started | 14 | 15
Completed | 13 | 15
Not Completed | 1 | 0
Not completed — Imperceptible tinnitus on the day of the assessment | 1 | 0

BASELINE CHARACTERISTICS:
Population: Thirty-three patients responded and attended the initial appointment, one was excluded for having only pulsatile tinnitus on the day of the appointment.
  Thirty-two patients started the study, being divided into study group (n=16) or placebo (n=16) through randomization. Each patient was their own control because this was a crossover study with an interval of 15 days between each evaluation.
Groups:
- Lidocaine 10%, Then Placebo: Lidocaine 10 MG/ML: Application of 10% topical lidocaine in the external auditory canal of tinnitus patients.
  The patient is instructed to lie down in lateral decubitus, with the ear in study facing upwards and 10% lidocaine is applied to the external auditory canal, using an eyedropper, until its complete filling (approximate average of 2ml).
  After an interval of 15 days the same procedure was done with placebo.
- Placebo, Then Lidocaine 10%: Distilled water: Application of distilled water in the external auditory canal of tinnitus patients.
  The patient is instructed to lie down in lateral decubitus, with the ear in study facing upwards and distilled water is applied to the external auditory canal, using an eyedropper, until its complete filling (approximate average of 2ml).
  After an interval of 15 days the same procedure was done with lidocaine.
- Total: Total of all reporting groups
Arm/Group | Lidocaine 10%, Then Placebo | Placebo, Then Lidocaine 10% | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.4 (14.22) | 55.5 (13.06) | 54 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 19
  Male | 5 | 8 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 16 | 32
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Brazil | 16 | 16 | 32
Tinnitus Handicap Inventory Score [Mean (Standard Deviation); unit: units on a scale] — The Tinnitus Handicap Inventory (THI) is a valuable self-report measure used to assess perceived tinnitus handicap severity. It consists of 25 items grouped into three subscales: functional, emotional, and catastrophic.
  The THI total score ranges from 0 to 100, with higher scores indicating greater tinnitus handicap severity. Very mild (score 0-16), Mild (score 18-36), Moderate (score 38-56), Severe (score 58-76), Catastrophic (score 78-100)
  units on a scale | 33.87 (21.31) | 29.25 (13.06) | 31.4 (17.1)
Study ear side right [Number; unit: participants] | 6 | 6 | 12
Presence of pain [Count of Participants; unit: Participants] | 6 | 7 | 13
Dizziness [Count of Participants; unit: Participants] | 3 | 3 | 6
Diabetes [Count of Participants; unit: Participants] | 2 | 2 | 4
Systemic arterial hypertension [Count of Participants; unit: Participants] | 7 | 3 | 10
Dyslipidemia [Count of Participants; unit: Participants] | 7 | 7 | 14
Hypothyroidism [Count of Participants; unit: Participants] | 1 | 1 | 2
Anxiety/Depression [Count of Participants; unit: Participants] | 7 | 6 | 13
Cervical spina dysfunction [Count of Participants; unit: Participants] — Cervical dysfunction was considered when the patient reported neck pain associated with image changes on cervical tomography or cervical magnetic resonance imaging.
  The measure used for this assessment was the presence (yes) or absence (no) of this type of dysfunction.
  Participants | 6 | 9 | 15
Bruxism/temporomandibular dysfunction [Count of Participants; unit: Participants] — Bruxism refers to the habit of grinding or clenching one's teeth, often unconsciously. It can occur during the day (awake bruxism) or at night (sleep bruxism). Temporomandibular dysfunction (TMD), on the other hand, encompasses a range of symptoms related to the temporomandibular joint (TMJ) and the surrounding muscles. These symptoms may include jaw pain, clicking, limited mouth opening, and headaches. We considered the patient's self-report as positive bruxism and as positive temporomandibular disorder when there was a diagnosis confirmed by a dentist.
  Participants | 9 | 9 | 18
Study ear side left [Count of Participants; unit: Participants] | 10 | 10 | 20
Presence of hearing loss [Count of Participants; unit: Participants] | 3 | 3 | 6
Somatosensory tinnitus [Count of Participants; unit: Participants] — Somatosensory tinnitus was considered positive when the following three conditions were present: tinnitus modulation through voluntary movements, somatic maneuvers, or tinnitus manipulation; onset of tinnitus associated with head and neck trauma or the onset of pain in the head and neck region; tinnitus accompanied by frequent neck pain, the presence of trigger points, the presence of muscle tension, temporomandibular disorder, or bruxism.
  Participants | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Change in Visual Analogue Scale (VAS) Score
Description: scale ranging from 0 to 10 points used to measure the intensity of tinnitus, where zero corresponds to the absence of tinnitus perception and 10 corresponds to the largest volume that the patient imagines that tinnitus may have.
Time Frame: Immediately before and 5 minutes after receiving intervention on days 1 and 15
Population: The mean VAS was compared between lidocaine and the placebo before and after the administration of each substance to evaluate the effect of lidocaine on tinnitus.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lidocaine 10% | Placebo
Number analyzed (Participants) | 31 | 29
score on a scale
  VAS before the application of the substances | 6.3 (1.8) | 6.3 (2.0)
  VAS after the application of the substances | 5.5 (2.1) | 5.2 (2.6)
Statistical Analysis 1: Comparison: Lidocaine 10% vs Placebo; The alternative hypothesis of this study is that 10% lidocaine, applied topically to the external auditory canal (EAC), acts on tinnitus intensity differently than placebo, while the null hypothesis is that there is no difference between the action of lidocaine and placebo on tinnitus intensity. The analyses were performed using the IBM-SPSS for Windows software version 22.0 and tabulated using the Microsoft-Excel 2010 software, and the tests were performed with a significance level of 5%; Test type: Other — VAS was described with the use of summary measures, and the variations between the applied substances were compared with the use of Generalized Estimating Equations (GEE) with normal marginal distribution and identity binding function, assuming an interchangeable correlation matrix between the substances (McCullagh; Nelder, 1989); Generalized Estimating Equations; VAS was described with the use of summary measures, and the variations between the applied substances were compared with the use of Generalized Estimating Equations (GEE) with normal marginal distribution and identity binding function, assuming an interchangeable correlation matrix between the substances (McCullagh; Nelder, 1989)

2. Primary Outcome: Change in Tinnitus Loudness
Description: Acuphenometry is a psychoacoustic test performed in an audiometry booth to measure tinnitus intensity. By comparing the intensity of tinnitus with the intensity sounds offered by the researcher, the tinnitus loudness is defined.
  Tinnitus loudness is measured in decibels and the higher the value found, the louder the tinnitus intensity.
Time Frame: Immediately before and 5 minutes after receiving intervention on days 1 and 15
Population: The mean Tinnitus loudness (decibels) was compared between lidocaine and the placebo before and after the administration of each substance to evaluate the effect of lidocaine on tinnitus.
Measure: Mean (Standard Deviation); unit: decibels
Arm/Group | Lidocaine 10% | Placebo
Number analyzed (Participants) | 31 | 29
decibels
  Tinnitus loudness before application of substances | 7.2 (7.8) | 6.4 (8.4)
  Tinnitus loudness after application of substances | 5.6 (7.7) | 4.6 (8.3)
Statistical Analysis 1: Comparison: Lidocaine 10% vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other — Tinnitus loudness was described with the use of summary measures, and the variations between the applied substances were compared with the use of Generalized Estimating Equations (GEE) with normal marginal distribution and identity binding function, assuming an interchangeable correlation matrix between the substances (McCullagh; Nelder, 1989); Tinnitus loudness was described with the use of summary measures, and the variations between the applied substances were compared with the use of Generalized Estimating Equations (GEE) with normal marginal distribution and identity binding function, assuming an interchangeable correlation matrix between the substances (McCullagh; Nelder, 1989)

3. Primary Outcome: Change in Minimum Masking Level (MML)
Description: Acuphenometry is a psychoacoustic test performed in an audiometry booth to measure minimum masking level. By comparing the intensity of tinnitus with the intensity sounds offered by the researcher, the minimum stimulus that masks tinnitus is determined.
  The minimum masking level is the intensity that an external sound must have to cover up tinnitus until it is no longer perceived by the patient. MML is measured in decibels.
  The lower the MML value, the more easily tinnitus can be masked, suggesting a lower degree of discomfort for the patient.
Time Frame: Immediately before and 5 minutes after receiving intervention on days 1 and 15
Population: The mean MML (decibels) was compared between lidocaine and the placebo before and after the administration of each substance to evaluate the effect of lidocaine on tinnitus.
Measure: Mean (Standard Deviation); unit: decibels
Arm/Group | Lidocaine 10% | Placebo
Number analyzed (Participants) | 31 | 29
decibels
  MML before the application of the substances | 4 (3) | 4.8 (2.4)
  MML after the application of the substances | 3.7 (2.9) | 3.8 (2.2)
Statistical Analysis 1: Comparison: Lidocaine 10% vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other — MML was described with the use of summary measures, and the variations between the applied substances were compared with the use of Generalized Estimating Equations (GEE) with normal marginal distribution and identity binding function, assuming an interchangeable correlation matrix between the substances (McCullagh; Nelder, 1989); MML was described with the use of summary measures, and the variations between the applied substances were compared with the use of Generalized Estimating Equations (GEE) with normal marginal distribution and identity binding function, assuming an interchangeable correlation matrix between the substances (McCullagh; Nelder, 1989)

ADVERSE EVENTS:
Time Frame: The adverse effects were collected up to 1 week after each intervention.
Arm/Group | Lidocaine 10% | Placebo
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/29
Other Adverse Events (participants affected / at risk) | 0/31 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-04): https://cdn.clinicaltrials.gov/large-docs/41/NCT05711641/Prot_SAP_000.pdf